CLINICAL TRIAL: NCT06922617
Title: Evaluating a Tobacco Harm Reduction Strategy Among Clients Enrolled in Substance Use Disorder Treatment
Brief Title: STEPS: Substance Use Trial of E-cigarettes or Pharmacotherapy for Smoking
Acronym: STEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin McClure, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00136062
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use; Substance Use Disorders
MeSH Terms: conditions — Tobacco Use; Substance-Related Disorders | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication (Experimental): This arm includes participants randomly assigned to the medication group. Participants will receive combination nicotine replacement therapy (NRT). The NRT will consist of transdermal patches and nicotine lozenges. Participants will receive study product for 12 weeks.
  Interventions: Drug: Quitting using Medication; Behavioral: Counseling
- Switching to an E-Cigarette (Experimental): This arm includes participants randomly assigned to the E-Cigarette Group. Participants will receive a study-provided e-cigarette product for 12 weeks.
  Interventions: Behavioral: Switching to E-Cigarette; Behavioral: Counseling

INTERVENTIONS:
Behavioral: Switching to E-Cigarette — Participants will receive twelve weeks of e-cigarette products with instructions to switch completely at switch date
  Arms: Switching to an E-Cigarette
Drug: Quitting using Medication — Participants will receive twelve weeks of FDA approved medication, combination NRT, with instructions to quit smoking cigarettes at quit date
  Arms: Medication
Behavioral: Counseling — Participants will recieve brief weekly counseling to support their quit or switch attempt from cigarettes.

SUMMARY:
The purpose of this study is to investigate whether non-cigarette tobacco products, namely e-cigarettes (nicotine vapes), can help people who smoke and are in treatment for substance use disorder quit smoking by switching completely to e-cigarettes as compared to FDA-approved medications, namely nicotine replacement therapy in the form of patches and lozenges. Participation will last 6 months and will include five in-person study visits and eleven virtual assessments. Participants will also complete a short daily diary on their phones each day for the first twelve weeks. To qualify, participants must be within 30 days of SUD treatment program admission. This study is being conducted at three outpatient SUD treatment programs across South Carolina. These sites include: 1) the Center for Drug and Alcohol Problems (CDAP) in Charleston, SC, 2) Behavioral Health Services of Pickens County (BHSPC) in Pickens, SC, and 3) Shoreline Behavioral Health Services in Conway, SC. the Medical University of South Carolina in Charleston, SC, Behavioral Health Services in Pickens, SC, and the Medical University of South Carolina in Florence, SC.

DETAILED DESCRIPTION:
Tobacco use rates among those with substance use disorders (SUD) are disproportionately high compared to the general population. While rates of tobacco use continue to decline in the general population, use rates among those with SUD have remained stagnant, with only slight declines noted in recent years. Despite this, clients enrolled in SUD treatment rarely engage in evidence-based tobacco treatment and many do not quit using tobacco during treatment. Continued tobacco use during SUD treatment results in worse substance-related treatment outcomes, as well as premature morbidity and mortality. Yet, surprisingly few rigorous randomized controlled trials (RCT) have been conducted to assess tobacco cessation in this population. Strategies to reduce the harmful effects of continued tobacco use in a SUD treatment population are urgently needed.

Importantly, those in SUD treatment who smoke cigarettes endorse an interest in quitting smoking, but quit rates are lower among a SUD population compared to the general population by about half. For example, within our own hospital system at the Medical University of South Carolina (MUSC), which employs an opt-out tobacco cessation approach for all inpatients, those with mental health diagnoses, including SUD, were less likely to report tobacco abstinence at 30-day follow-up post-discharge, compared to those without mental health diagnoses. There is a clear public health need to address the harmful impact of combustible tobacco use among those enrolled in treatment for SUD and ensure that these strategies, should they be efficacious in reducing harm, are acceptable and feasible for SUD clients, program staff and leadership. The need to address combustible tobacco use in this population has been present for decades and yet advances in this area have been minimal. Those in SUD treatment are still disproportionately impacted by the harms of combustible tobacco, which may be due, in large part, to the barriers that exist in treating tobacco as part of SUD standard of care.

Participants will be randomized 1:1 to: 1) switch exclusively to ENDS, or 2) quit tobacco with NRT. The aims of this study are to: 1) evaluate if switching to ENDS leads to greater rates of 7-day biologically confirmed point prevalence abstinence (PPA) from cigarette smoking at 12 weeks compared to quitting with NRT among those enrolled in SUD treatment (Aim 1), 2) evaluate patient, provider, and organizational-level implementation outcomes using mixed methods according to the Proctor framework, which describes barriers and facilitators of successful implementation of an intervention (Aim 2), and 3) assess the impact of switching to ENDS compared to quitting with NRT on SUD treatment outcomes and engagement to test for non-inferiority over 12 weeks (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

1. 21+ years of age,
2. smoke at least 5 cigarettes per day daily or near daily for the past 6 months,
3. be within 90 days of the first outpatient SUD treatment session and have an active SUD diagnosis,
4. must submit a breath CO sample of ≥ 7 parts per million at screening and a positive instant-read urinary cotinine test,
5. have had at least one failed smoking quit attempt in their lifetime,
6. have interest in reducing smoking, quitting smoking, or switching to a less harmful product, and
7. if female, agrees to use a form of birth control during the study.

Exclusion Criteria:

1. any significant or unstable medical or psychiatric concern that would affect safety,
2. current use of pharmacotherapy with smoking cessation efficacy,
3. pregnant, breastfeeding, or trying to become pregnant,
4. contraindicated for NRT, and
5. currently using an ENDS on 10+ days out of the past 30.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Abstinence from smoking at end of treatment | 7 days
  7-day biologically confirmed point prevelance abstinence from cigarette smoking at Week 12 end of treatment visit

SECONDARY OUTCOMES:
Acceptability of the intervention | 12 weeks
  4-item Acceptability of the Intervention Measure where higher scores indicate greater acceptability (range 1-5)
Number of negative urine drug screens | 12 weeks
  Number of negative urine drug screens (for the primary substance of use) submitted during the 12 week treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - MUSC Charleston, Center for Drug and Alcohol Problems, Charleston, South Carolina
  - Shoreline Behavioral Health Services, Conway, South Carolina
  - Behavioral Health Services of Pickens County, Pickens, South Carolina